CLINICAL TRIAL: NCT03476408
Title: Investigation of the Relationship Between Plantar Sensation, Balance, Risk of Falling and Gait in Patients With Schizophrenia
Brief Title: Plantar Sensation, Balance, Risk of Falling and Gait in Patients With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Caner Karartı, Principal Investigator, Hacettepe University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2018100
Record Dates: First submitted 2018-03-15; First posted 2018-03-26 (Actual); Last update posted 2018-03-26 (Actual); Status verified 2018-03

CONDITIONS: Plantar Sensation; Balance; Distorted; Fall; Gait Disorders, Neurologic
MeSH Terms: conditions — Gait Disorders, Neurologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Group Correlation (Experimental): Correlation between these topics.
  Interventions: Other: Correlation / Observational

INTERVENTIONS:
Other: Correlation / Observational — correlation between Plantar Sensation, Balance, Risk of Falling and Gait in Patients With Schizophrenia

SUMMARY:
Cerebellar vermis anomalies are present in schizophrenic individuals. This condition leads to postural balance problems. Foot and ankle complex have a special role for maintaining balance. However, there is no study about this topic in schizophrenic individuals.

ELIGIBILITY:
Inclusion Criteria:

* diagnose of schizophrenia according to DSM-5
* being an individual in remission against the risk of having an attack
* individuals who use the same psychotropic drugs for at least 4 weeks

Exclusion Criteria:

* Individuals with physical and neurological comorbidities

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2018-03-15 (Actual); Study Completion 2018-03-15 (Actual)

PRIMARY OUTCOMES:
Semmes-Weinstein Monofilament test | 1 year
  Plantar sensation
Berg Balance Scale | 1 year
  Balance
Tinetti Fall Risk Scale | 1 year
  Risk of Falling
Spinal Mouse | 1 year
  Spinal flexibility for balance
Walk a Line Battery | 1 year
  Gait

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Ahi Evran University, Kırşehir, Kirşehi̇r
  - Ahi Evran University, Kırşehir

IPD SHARING:
Plan to Share IPD: Undecided